CLINICAL TRIAL: NCT00658879
Title: SPECIAL INVESTIGATION OF SOMAVERT -LONG TERM USE-
Brief Title: Long Term Use of Somavert (Pegvisomant) For A Regulatory Post Marketing Commitment Plan
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6291023
Record Dates: First submitted 2008-04-09; First posted 2008-04-15 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-08

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — pegvisomant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Somavert (Pegvisomant): Patients taking Somavert (Pegvisomant).
  Interventions: Drug: Somavert (Pegvisomant)

INTERVENTIONS:
Drug: Somavert (Pegvisomant) — Somavert (Pegvisomant) 10, 15 or 20mg powder and solvent for solution for injection.
  Dosage, Frequency : According to Japanese LPD.
  Duration : According to the protocol of A6291023, the duration of the investigation for findings regarding safety and efficacy of a patient is from the first drug administration to the 5 years after the first administration.

SUMMARY:
The objective of this surveillance is to collect information about 1) adverse drug reaction not expected from the LPD (unknown adverse drug reaction), 2) the incidence of adverse drug reactions in this surveillance, and 3)factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first Somavert (Pegvisomant) should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

Patients need to be administered Somavert (Pegvisomant) in order to be enrolled in the surveillance.

Exclusion Criteria:

Patients not administered Somavert (Pegvisomant).

Min Age: 0 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A6291023 prescribes Somavert (Pegvisomant).
Sampling Method: Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2007-08-07 (Actual); Primary Completion 2016-11-09 (Actual); Study Completion 2016-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6291023&StudyName=Long%20Term%20Use%20of%20Pegvisomant%20For%20A%20Regulatory%20Post%20Marketing%20Commitment%20Plan%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Somavert (Pegvisomant): Participants who received Somavert as indicated in the approved local product document were observed for a period of 5 years. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | Somavert (Pegvisomant)
Started | 251
Completed | 250
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: A total of 251 participants were enrolled in this study. Of the 251 participants, 1 participant was excluded from the baseline analysis due to protocol violation.
Arm/Group | Somavert (Pegvisomant)
Number analyzed (Participants) | 250
Age, Customized [Number; unit: Participants]
  <15 years | 2
  ≥15 and <65 years | 198
  ≥65 years | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141
  Male | 109
Hepatic Function Disorder [Number; unit: Participants]
  Absent | 234
  Present | 16
Renal Impairment [Number; unit: Participants]
  Absent | 241
  Present | 9
Diabetes Mellitus (Concurrent Disease) [Number; unit: Participants]
  Absent | 139
  Present | 111

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Somavert in a participant who received Somavert. A treatment-related serious adverse event was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to Somavert was assessed by the physician.
Time Frame: 5 years
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and had received Somavert at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Somavert (Pegvisomant)
Number analyzed (Participants) | 250
Participants
  Treatment-related Adverse Event | 89
  Treatment-related Serious Adverse Event | 20

2. Primary Outcome: Number of Participants With Treatment-Related Adverse Events Unexpected From Japanese Package Insert
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Somavert in a participant who received Somavert. Expectedness of the adverse event was determined according to the Japanese package insert. Relatedness to Somavert was assessed by the physician.
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Somavert (Pegvisomant)
Number analyzed (Participants) | 250
Participants | 9

3. Primary Outcome: Number of Participants With Treatment-Related Adverse Events by Gender
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Somavert in a participant who received Somavert. Relatedness to Somavert was assessed by the physician. Participants with treatment-related adverse events were counted by gender to assess whether it was a risk factor for the occurrence of treatment-related adverse events.
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Somavert (Pegvisomant)
Number analyzed (Participants) | 250
Participants
  Female: number analyzed (Participants) | 141
  Female | 52
  Male: number analyzed (Participants) | 109
  Male | 37

4. Primary Outcome: Number of Participants With Treatment-Related Adverse Events by Age
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Somavert in a participant who received Somavert. Relatedness to Somavert was assessed by the physician. Participants with treatment-related adverse events were counted by age to assess whether it was a risk factor for the occurrence of treatment-related adverse events.
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Somavert (Pegvisomant)
Number analyzed (Participants) | 250
Participants
  <15 years: number analyzed (Participants) | 2
  <15 years | 2
  ≥15 and <65 years: number analyzed (Participants) | 198
  ≥15 and <65 years | 75
  ≥65 years: number analyzed (Participants) | 50
  ≥65 years | 12

5. Primary Outcome: Number of Participants With Treatment-Related Adverse Events for Participants With Hepatic Function Disorder
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Somavert in a participant who received Somavert. Relatedness to Somavert was assessed by the physician. Participants with treatment-related adverse events were counted by hepatic function disorder to assess whether it was a risk factor for the occurrence of treatment-related adverse events.
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Somavert (Pegvisomant)
Number analyzed (Participants) | 250
Participants
  Without hepatic function disorder: number analyzed (Participants) | 234
  Without hepatic function disorder | 85
  With hepatic function disorder: number analyzed (Participants) | 16
  With hepatic function disorder | 4

6. Primary Outcome: Number of Participants With Treatment-Related Adverse Events for Participants With Renal Impairment
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Somavert in a participant who received Somavert. Relatedness to Somavert was assessed by the physician. Participants with treatment-related adverse events were counted by renal impairment to assess whether it was a risk factor for the occurrence of treatment-related adverse events.
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Somavert (Pegvisomant)
Number analyzed (Participants) | 250
Participants
  Without renal impairment: number analyzed (Participants) | 241
  Without renal impairment | 88
  With renal impairment: number analyzed (Participants) | 9
  With renal impairment | 1

7. Primary Outcome: Number of Participants With Treatment-Related Adverse Events for Participants With Diabetes Mellitus (Concurrent Disease)
Description: A treatment-related adverse event was any untoward medical occurrence attributed to Somavert in a participant who received Somavert. Relatedness to Somavert was assessed by the physician. Participants with treatment-related adverse events were counted by diabetes mellitus (concurrent disease) to assess whether it was a risk factor for the occurrence of treatment-related adverse events.
Time Frame: 5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Somavert (Pegvisomant)
Number analyzed (Participants) | 250
Participants
  Without diabetes mellitus: number analyzed (Participants) | 139
  Without diabetes mellitus | 57
  With diabetes mellitus: number analyzed (Participants) | 111
  With diabetes mellitus | 32

8. Primary Outcome: Clinical Effectiveness Rate
Description: Clinical effectiveness rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of assessable effectiveness analysis population, was presented. Clinical effectiveness of Somavert was assessed as "effective," "ineffective" or "unassessable" by the physician. Overall effectiveness of Somavert was determined by the physician based on clinical symptoms, laboratory values, and other examinations such as ring size.
Time Frame: 5 years
Population: The efficacy analysis set comprised of participants in the safety analysis set who had effectiveness evaluation (overall evaluation by the physician based upon change in clinical symptoms and laboratory findings) at least once. Participants evaluated as "unassessable" were excluded from the calculation.
Measure: Number; unit: Percentage of Participants
Arm/Group | Somavert (Pegvisomant)
Number analyzed (Participants) | 225
Percentage of Participants | 96.4

9. Primary Outcome: Clinical Effectiveness Rate by Gender
Description: Clinical effectiveness rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of assessable effectiveness analysis population, was presented. Clinical effectiveness of Somavert was assessed as "effective," "ineffective" or "unassessable" by the physician. Overall effectiveness of Somavert was determined by the physician based on clinical symptoms, laboratory values, and other examinations such as ring size. Participants achieved clinical effectiveness by gender were counted to assess whether it contributes to the clinical effectiveness.
Time Frame: 5 years
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | Somavert (Pegvisomant)
Number analyzed (Participants) | 225
Percentage of Participants
  Female: number analyzed (Participants) | 126
  Female | 96.8
  Male: number analyzed (Participants) | 99
  Male | 96.0

10. Primary Outcome: Clinical Effectiveness Rate by Age
Description: Clinical effectiveness rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of assessable effectiveness analysis population, was presented. Clinical effectiveness of Somavert was assessed as "effective," "ineffective" or "unassessable" by the physician. Overall effectiveness of Somavert was determined by the physician based on clinical symptoms, laboratory values, and other examinations such as ring size. Participants achieved clinical effectiveness by age were counted to assess whether it contributes to the clinical effectiveness.
Time Frame: 5 years
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | Somavert (Pegvisomant)
Number analyzed (Participants) | 225
Percentage of Participants
  <15 years: number analyzed (Participants) | 2
  <15 years | 50.0
  ≥15 and <65 years: number analyzed (Participants) | 180
  ≥15 and <65 years | 96.1
  ≥65 years: number analyzed (Participants) | 43
  ≥65 years | 100.0

11. Primary Outcome: Clinical Effectiveness Rate in Participants With Hepatic Function Disorder
Description: Clinical effectiveness rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of assessable effectiveness analysis population, was presented. Clinical effectiveness of Somavert was assessed as "effective," "ineffective" or "unassessable" by the physician. Overall effectiveness of Somavert was determined by the physician based on clinical symptoms, laboratory values, and other examinations such as ring size. Participants achieved clinical effectiveness by hepatic function disorder were counted to assess whether it contributes to the clinical effectiveness.
Time Frame: 5 years
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | Somavert (Pegvisomant)
Number analyzed (Participants) | 225
Percentage of Participants
  Without hepatic function disorder: number analyzed (Participants) | 212
  Without hepatic function disorder | 96.7
  With hepatic function disorder: number analyzed (Participants) | 13
  With hepatic function disorder | 92.3

12. Primary Outcome: Clinical Effectiveness Rate in Participants With Diabetes Mellitus (Concurrent Disease)
Description: Clinical effectiveness rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of assessable effectiveness analysis population, was presented. Clinical effectiveness of Somavert was assessed as "effective," "ineffective" or "unassessable" by the physician. Overall effectiveness of Somavert was determined by the physician based on clinical symptoms, laboratory values, and other examinations such as ring size. Participants achieved clinical effectiveness by diabetes mellitus (concurrent disease) were counted to assess whether it contributes to the clinical effectiveness.
Time Frame: 5 years
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | Somavert (Pegvisomant)
Number analyzed (Participants) | 225
Percentage of Participants
  Without diabetes mellitus: number analyzed (Participants) | 126
  Without diabetes mellitus | 96.0
  With diabetes mellitus: number analyzed (Participants) | 99
  With diabetes mellitus | 97.0

ADVERSE EVENTS:
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as non-serious in another subject, or one subject may have experienced both serious and non-serious events during the study.
Arm/Group | Somavert (Pegvisomant)
Serious Adverse Events (participants affected / at risk) | 39/250
Other Adverse Events (participants affected / at risk) | 117/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Somavert (Pegvisomant) (N=250)
Appendicitis (Infections and infestations) | 1
Cholecystitis infective (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Pituitary tumour recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Contrast media allergy (Immune system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Hypopituitarism (Endocrine disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Altered state of consciousness (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Aortic valve incompetence (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 2
Large intestine polyp (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Volvulus (Gastrointestinal disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Condition aggravated (General disorders) | 2
Disease progression (General disorders) | 11
Malaise (General disorders) | 1
Platelet count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Cardiac resynchronisation therapy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Somavert (Pegvisomant) (N=250)
Anaemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Deafness unilateral (Ear and labyrinth disorders) | 1
Dry eye (Eye disorders) | 1
Eyelid ptosis (Eye disorders) | 1
Iritis (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 3
Large intestine polyp (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 1
Condition aggravated (General disorders) | 2
Disease progression (General disorders) | 5
Facial pain (General disorders) | 1
Fatigue (General disorders) | 1
Induration (General disorders) | 1
Injection site erythema (General disorders) | 2
Injection site hypertrophy (General disorders) | 3
Injection site induration (General disorders) | 4
Injection site pain (General disorders) | 1
Injection site pruritus (General disorders) | 3
Injection site swelling (General disorders) | 2
Malaise (General disorders) | 4
Alcoholic liver disease (Hepatobiliary disorders) | 2
Cholangitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 33
Hepatic steatosis (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 5
Bronchitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood glucose increased (Investigations) | 6
Blood growth hormone increased (Investigations) | 4
Blood pressure increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 6
Glycosylated haemoglobin increased (Investigations) | 3
Insulin-like growth factor increased (Investigations) | 2
Liver function test abnormal (Investigations) | 2
Low density lipoprotein increased (Investigations) | 1
Weight increased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 7
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 3
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Hyperlipidaemia (Metabolism and nutrition disorders) | 2
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Obesity (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Joint lock (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Pituitary tumour recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Diabetic neuropathy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 9
Memory impairment (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Renal tubular acidosis (Renal and urinary disorders) | 1
Ureteric stenosis (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.